CLINICAL TRIAL: NCT01249547
Title: Phase 2 Study of Axitinib in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Nasopharyngeal Carcinoma (NPC) Axitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC022
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Recurrent or Metastatic NPC
MeSH Terms: conditions — Recurrence | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axitinib arm (Experimental)
  Interventions: Drug: axitinib

INTERVENTIONS:
Drug: axitinib — starting dose of 5 mg twice daily for 4 consecutive weeks without interruption.

SUMMARY:
This is an open-label, single arm, phase 2 clinical trial evaluating the activity and safety of single-agent axitinib in recurrent or metastatic NPC patients who failed at least one line of platinum based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of nasopharyngeal carcinoma (NPC) (either at initial diagnosis or at recurrence).
* Patients with recurrent or metastatic NPC that has progressed following one line of prior platinum-based chemotherapy.
* Disease must be not amenable to potentially curative radiotherapy or surgery.
* Measurable disease according to RECIST.
* Age 18 or above; ECOG performance 0 or 1.
* Adequate bone marrow, renal and hepatic reserve.

Exclusion Criteria:

* Presence of local recurrence
* Presence of neck lymph node recurrence invading vascular structure;
* Presence of central lung lesions involving major blood vessels;
* History of hemoptysis or epistaxis within 4 weeks;
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite adequate medical therapy;
* Gastrointestinal abnormalities, including inability to take oral medication or malabsorption syndrome;
* Concurrent use or anticipated need for treatment with known potent CYP3A4 inhibitors or CYP3A4 /CYP1A2 inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (clinical benefit rate) of single-agent axitinib in patients with recurrent or metastatic NPC, and its impact on disease progression. | 3 years

SECONDARY OUTCOMES:
To assess objective response rate | 3 years
To assess duration of response | 3 years
To assess progression-free survival | 3 Years
To assess overall survival | 3 Years
To evaluate the safety and tolerability of axitinib | 3 years
To evaluate axitinib plasma pharmacokinetics and to correlate these plasma concentrations with efficacy and safety parameters | 3 years
To study blood and tissue biomarkers and correlate with cancer- and treatment-related outcomes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony TC Chan, MD, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong